CLINICAL TRIAL: NCT04818463
Title: Characterization and Verification of the Intensive Care Standard Operating Procedure (SOP) Adherence of the Treated COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: QUALITY COVID-19
Record Dates: First submitted 2021-03-18; First posted 2021-03-26 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As part of the internal quality management (QM project), this retrospective cohort study examines the adherence to Standard Operating Procedures (SOP) of the COVID-19 patients treated since January 1st, 2020 to February 28th, 2021 in intensive care units of the Clinic for Anesthesiology m.S. operative intensive care medicine CCM / CVK.

ELIGIBILITY:
Inclusion Criteria:

* During the intensive care stay with SARS-CoV-2 infected intensive care patients of the Charité - Universitätsmedizin Berlin, admitted to the intensive care units of the Department of Anesthesiology and operative intensive care medicine (CCM / CVK)
* Treatment period: 01/01/2020 to 02/28/2021
* At least 18 years old

Exclusion Criteria:

• Incomplete electronic documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the intensive care stay with SARS-CoV-2 infected intensive care adult patients
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
SOP "Analgesia, sedation, delirium and pain therapy" | 01.01.2020 - 28.02.2021
  SOP adherence to the selected SOP "Analgesia, sedation, delirium and pain therapy". Process: daily implementation yes / no - yes> 70%

SECONDARY OUTCOMES:
SOP "Treatment of acute respiratory distress syndrome (ARDS)" | 01.01.2020 - 28.02.2021
  SOP adherence to the selected SOP "Treatment of acute respiratory distress syndrome (ARDS)" Process: daily implementation yes / no - yes> 70%
SOP "Infectious treatment" | 01.01.2020 - 28.02.2021
  SOP adherence to the selected SOP "Infectious treatment" Process: daily implementation yes / no - yes> 70%
SOP "Weaning" | 01.01.2020 - 28.02.2021
  SOP adherence to the selected SOP "Weaning"
SOP "Nutrition" | 01.01.2020 - 28.02.2021
  SOP adherence to the selected SOP "Nutrition" Process: daily implementation yes / no - yes> 70%
SOP "Sepsis" | 01.01.2020 - 28.02.2021
  SOP adherence to the selected SOP "Sepsis" Process: daily implementation yes / no - yes> 70%

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Campus Virchow-Klinikum, Berlin, Germany